CLINICAL TRIAL: NCT00217399
Title: A Phase I/II Trial of BAY 43-9006 (Sorafenib) in Combination With Anastrozole in Patients With Metastatic Breast Cancer
Brief Title: Sorafenib and Anastrozole in Treating Postmenopausal Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00069; NCI-2009-00069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000440067; 2004-251; 2004-251 (Other: Lombardi Comprehensive Cancer Center at Georgetown University); 6584 (Other: CTEP)
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Results first posted 2013-02-12 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Sorafenib; Anastrozole

ARMS (1):
- Treatment (Experimental): PHASE I: Patients receive oral sorafenib twice daily and oral anastrozole once daily on days 1-28.
  Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 patients are treated at the MTD.
  PHASE II: Patients receive sorafenib at the MTD and anastrozole as in phase I.
  Interventions: Drug: sorafenib tosylate; Drug: anastrozole

INTERVENTIONS:
Drug: sorafenib tosylate — Given orally
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Drug: anastrozole — Given orally
  Other Names: ANAS; Arimidex; ICI-D1033

SUMMARY:
Sorafenib may stop the growth of tumor cells by blocking blood flow to the tumor and by blocking some of the enzymes needed for cell growth. Estradiol can cause the growth of breast cancer. Hormone therapy using anastrozole may fight breast cancer by blocking the use of estradiol by the tumor cells. Sometimes when hormone therapy is given, it does not stop the growth of tumor cells. The tumor is said to be resistant to hormone therapy. Giving sorafenib together with anastrozole may reduce drug resistance and allow the tumor cells to be killed. This phase I/II trial is studying the side effects and best dose of sorafenib when given in combination with anastrozole and to see how well they work in treating postmenopausal women with metastatic breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the clinical benefit rate of sorafenib in combination with anastrazole in women with estrogen receptor- and/or progesterone receptor-positive metastatic breast cancer.

II. Determine the recommended phase II dose of sorafenib when administered with anastrozole in these patients.

SECONDARY OBJECTIVES:

I. Determine the toxic effects of this regimen in these patients. II. Determine the changes in Raf-MAPK and VEGF-signaling pathways in tumor tissue and stroma before and after treatment with this regimen in these patients.

OUTLINE: This is a multicenter, dose-escalation study of sorafenib.

PHASE I: Patients receive oral sorafenib twice daily and oral anastrozole once daily on days 1-28.

Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of sorafenib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 patients are treated at the MTD.

PHASE II: Patients receive sorafenib at the MTD and anastrozole as in phase I.

After completion of study treatment, patients are followed every 4-8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer
* Metastatic disease
* Measurable disease, defined as >=1 unidimensionally measurable lesion, including >= 1 of the following:

  * Lesion >= 10 mm on CT scan (5 mm sections)
  * Lesion >= 20 mm on CT scan or MRI (10 mm sections)
  * Bone disease that is >= 10 mm on MRI
  * Lytic bone lesions that are >= 10 mm on CT scan (with 5 mm sections) OR >= 20 mm on plain film or CT scan (with 10 mm sections)
  * Lesion >= 10 mm on physical exam
* Patients must have received >= 1 prior aromatase inhibitor in either the adjuvant or metastatic setting and must have had either disease recurrence or disease progression on a prior aromatase inhibitor therapy
* No brain metastases diagnosed within the past 6 months OR previously untreated brain metastases
* Estrogen receptor-positive and/or progesterone receptor-positive, defined as > 1% staining by immunohistochemistry or > 10 fmol/mg of protein by radio-ligand dextran-coated steroid binding assay
* Postmenopausal, as defined by 1 of the following:

  * Prior bilateral oophorectomy
  * No menses for >= 12 months in patients with an intact uterus
  * Follicle-stimulating hormone (FSH) in postmenopausal range in patients < 60 years of age who have had a prior hysterectomy or have been amenorrheic for >= 3 months
  * Age >= 60 years
  * Pre- or perimenopausal patients receiving monthly injections of goserelin at a dose of 3.6 mg are eligible
* ECOG 0-2
* More than 3 months
* Absolute neutrophil count >= 1,500/mm3 Platelet count >= 100,000/mm3 No bleeding diathesis
* Bilirubin =< 1.5 times upper limit of normal (ULN AST and ALT =< 2.5 times ULN
* Systolic blood pressure (BP) < 150 mm Hg and diastolic BP < 100 mm Hg on at least one reading prior to study entry No uncontrolled hypertension
* None of the following within the past 6 months:

  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Myocardial infarction
  * Cardiac arrhythmia with hemodynamic compromise
* Not pregnant or nursing
* Able to swallow oral medication
* No known HIV positivity
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other active invasive malignancy within the past 5 years except nonmelanoma skin cancer or treated carcinoma in situ of the cervix
* No other uncontrolled illness
* More than 4 weeks since prior chemotherapy
* No more than 2 prior chemotherapy regimens for metastatic disease
* At least 8 weeks since prior anastrozole therapy
* Concurrent steroids allowed if dose is stable
* More than 4 weeks since prior radiotherapy
* More than 4 weeks since prior major surgery
* Recovered from prior therapy
* No prior sorafenib
* No concurrent therapeutic anticoagulation
* Concurrent prophylactic anticoagulation (i.e., low-dose warfarin) for venous or arterial access devices allowed provided PT and PTT are =< 1.5 times ULN
* No concurrent agents that may interact with sorafenib, including any of the following:

  * Hypericum perforatum (St. John's wort)
  * Rifampin
  * P450 CYP3A4 enzyme-inducing anticonvulsants (e.g., phenytoin, carbamazepine, or phenobarbital)
* No other concurrent investigational agents

Exclusion Criteria:

* estrogen receptor status unknown
* history of myocardial infarction within 6 months
* performance status 3
* performance status 4
* premenopausal
* progesterone receptor status unknown
* HIV positive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-06; Primary Completion 2009-07 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudine Isaacs, Principal Investigator — Lombardi Comprehensive Cancer Center at Georgetown University
Locations (1):
- Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 22-Sep-2005 through 01-Jul-2009
Groups:
- Sorafenib and Anastrozole: A single arm of 35 patients with advanced or metastatic breast cancer receiving a combination of sorafenib and anastrozole.
Period: Overall Study
Arm/Group | Sorafenib and Anastrozole
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib and Anastrozole
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Complete Response + Partial Response + Stable Disease > 24 Weeks
Description: Clinical Outcome measured using Response Evaluation Criteria In Solid Tumors (RECIST,)V1.0, and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), a tumor that is neither growing nor shrinking.
  A patient has clinical benefit from treatment if CR + PR + SD > 24 weeks.
Time Frame: 24 weeks
Population: Female patients with advanced or metastatic breast cancer. The protocol was initiated with intention to treat every patient enrolled with a sorafenib and anastrozole combination.
Measure: Number; unit: participants
Groups:
- Sorafenib and Anastrozole: All patients receive sorafenib and anastrozole.
Arm/Group | Sorafenib and Anastrozole
Number analyzed (Participants) | 35
participants | 35 [20 to 25]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of patients treated with the sorafenib / anastrozole combination who experienced Grade 1-4 adverse events according to NCI common terminology criteria for adverse events (CTCAE) version 3.0
Time Frame: 1 year
Population: All 35 patients enrolled in the study were assessed for adverse events according to NCI common terminology criteria for adverse events (CTCAE) version 3.0.
Measure: Number; unit: participants
Groups:
- Sorefenib and Anastrozole: All patients receive sorafenib (400mg by mouth twice daily) and anastrazole (1 mg by mouth daily)
Arm/Group | Sorefenib and Anastrozole
Number analyzed (Participants) | 35
participants | 35

3. Secondary Outcome: Tumor Marker Analysis
Description: Number of participants with significant change in the following circulating tumor biomarkers, measured by flow cytometry: cluster designation (CD)146, CD133. Values were normalized by CD45 values(ie CD146+/CD45- and CD133+/CD45-).
Time Frame: 1 year
Population: 14 subjects had blood specimens available for analysis
Measure: Number; unit: participants
Groups:
- Circulating Endothelial Cells: All patients received sorafenib and anastrozole. Blood was drawn prior to beginning treatment and at set time points to analyze for circulating endothelial cells by flow cytometry
Arm/Group | Circulating Endothelial Cells
Number analyzed (Participants) | 14
participants | 14

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Sorafenib and Anastrozole
Serious Adverse Events (participants affected / at risk) | 12/35
Other Adverse Events (participants affected / at risk) | 35/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib and Anastrozole (N=35)
hand-foot syndome (Skin and subcutaneous tissue disorders) | 12 (12)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib and Anastrozole (N=35)
Emesis (Gastrointestinal disorders) | 14 (14)
acne (Skin and subcutaneous tissue disorders) | 2 (2)
anorexia (Metabolism and nutrition disorders) | 11 (11)
anthralgias (Musculoskeletal and connective tissue disorders) | 9 (9)
dehydration (General disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 22 (22)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
elevated liver function tests (Hepatobiliary disorders) | 7 (7)
fatigue (General disorders) | 23 (23)
headache (General disorders) | 9 (9)
hypertension (Cardiac disorders) | 11 (11)
hypophosphatemia (General disorders) | 1 (1)
hypotension (Blood and lymphatic system disorders) | 2 (2)
infection (Infections and infestations) | 3 (3)
joint function (Musculoskeletal and connective tissue disorders) | 4 (4)
mucositis (General disorders) | 8 (8)
nausea (Gastrointestinal disorders) | 21 (21)
neutropenia (Blood and lymphatic system disorders) | 3 (3)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 17 (17)
rigors/chills (General disorders) | 5 (5)
thrombosis (Cardiac disorders) | 1 (1)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less